CLINICAL TRIAL: NCT05668182
Title: Early Outcomes Utilizing the TRUMATCH Graft Cage for Segmental Long Bone Defects: A Case Series
Brief Title: A Case Series: TRUMATCH Graft Cage for Segmental Long Bone Defects
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, William Kent, Assistant Professor of Orthopaedic Surgery, University of California, San Diego
Other Study IDs: 210671
Record Dates: First submitted 2022-12-19; First posted 2022-12-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Tibia Fracture; Humerus Fracture; Femoral Fracture; Long Bone Segmental Defect
MeSH Terms: conditions — Tibial Fractures; Humeral Fractures; Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: TRUMATCH Graft Cage — TRUMATCH Graft Cage for surgical repair of segmental long bone defect

SUMMARY:
This project consists of a prospective case design. Study candidates will include all patients ages 18 and over who were evaluated at UCSD and found to have a critical-sized humerus, femur, or tibia segmental defect that would be fixed through surgery. Patients who consent to study participation will receive the TRUMATCH Graft Cage for their long bone segmental defect repair. Data on healing rates, complication rates, re-operation rates, time to return to normal activity, and pain levels will be collected for each participation. After 3 years of data collection, we will analyze this data to provide further insight on the utility of the TRUMATCH Graft Cage. Given the significant difficulty with repairing segmental long bone defects, it is imperative to evaluate novel systems to appropriately manage these injuries.

ELIGIBILITY:
Inclusion Criteria:

* Humerus, femur, or tibia segmental defects requiring surgery
* Evaluation and treatment at UCSD
* Ages 18 year and older
* Abiltiy to understand the content of the patient information/informed consent form

Exclusion Criteria:

* Any not medically managed severe systemic disease
* Their doctor has decided that it is in the patient's best interest to receive a different method of repair
* Their doctor has determined that the patient has a condition that would make them unsuitable for participation in the study
* Pregnancy or women planning to conceive within the subject participation period (1 year) note: pregnancy will be self-reported and no test will be performed to test for it
* Prisoner
* Participation in any other pharmacologic or medicinal product study within the previous month that could influence the results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older presenting to UCSD Medical Center with a humerus, femur, or tibia segmental defects requiring surgery
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Use of the TRUMATCH Graft Cage- Long Bone | 2 years

SECONDARY OUTCOMES:
Healing Rates | 2 years
Reoperation Rates | 2 years
Complications | 2 years
Pain Scores | 2 years
Time to Return to Normal Activity | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States